CLINICAL TRIAL: NCT02428491
Title: Immunogenicity and Safety of Sanofi Pasteur's DTaP-IPV-Hep B-PRP-T Combined Vaccine Given as a Three-Dose Primary Series at 2, 3, and 4 Months of Age and Followed by a Booster Dose Given at 16 to 17 Months of Age in Vietnamese Infants Who Previously Received a Dose of Hepatitis B Vaccine at Birth or Within 1 Week After Birth
Brief Title: Immunogenicity and Safety of Sanofi Pasteur's Combined Vaccine Given as a Three-Dose Primary Series at 2, 3,4 Months of Age and Followed by a Booster Dose Given at 16 to 17 Months of Age in Vietnamese Infants Who Previously Received a Dose of Hepatitis B Vaccine at Birth or Within 1 Week After Birth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A3L35; U1111-1143-8177 (Other: WHO); NCT02821195 (obsolete NCT alias)
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Diphtheria; Tetanus; Pertussis; Poliomyelitis; Hepatitis B; Haemophilus Influenzae Type b
Keywords: Diphtheria; Tetanus; Pertussis; Poliomyelitis; Hepatitis B; Haemophilus Influenzae Type b; DTaP-IPV-Hep B-PRP-T Combined Vaccine (Hexaxim®)
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis; Hepatitis B; Haemophilus Infections | interventions — DTaP-IPV-HB-PRP-T vaccine

STUDY DESIGN:
Intervention Model Description: Participants in this trial were randomized in a 1:1 ratio in 2 cohorts. All participants in both cohorts received Sanofi Pasteur's DTaP-IPV-HB-PRP~T combined vaccine in a 3-dose Infant Series. Participants from Cohort 1 provided blood samples for immunogenicity assessment and were evaluated for safety and immunogenicity. Participants in Cohort 2 did not provide any blood samples for immunogenicity analysis and were evaluated for safety only.
Oversight: Data Monitoring Committee: No

ARMS (1):
- DTaP-IPV-HB-PRP~T Vaccine (Experimental): All participants will receive 3 doses of 0.5 mL DTaP-IPV-HB-PRP~T combined vaccine, intramuscularly, at 2, 3 and 4 months of age (primary series), followed by a booster dose approximately 12 months after the completion of the primary series (at 16 to 17 months of age).
  Interventions: Biological: Hexaxim®

INTERVENTIONS:
Biological: Hexaxim® — DTaP-IPV-Hep B-PRP-T combined vaccine, 0.5 mL, Intramuscular
  Other Names: Hexyon®; Hexacima®

SUMMARY:
The purpose of this study is to describe the immunogenicity and safety of Sanofi Pasteur's DTaP-IPV-Hep B-PRP-T fully liquid combined hexavalent vaccine (Hexaxim®) administered at 2, 3, and 4 months of age and at 16 to 17 months of age in infants and toddlers who received a dose of Hep B vaccine at birth or within 1 week after birth.

Primary Objective:

* To describe the safety profile after each and all doses of Sanofi-Pasteur's DTaP-IPV-Hep B-PRP-T combined vaccine in Vietnamese infants and toddlers.

Secondary Objective:

* To demonstrate the non-inferiority of the immune response to all antigens induced by the study vaccine in Vietnamese infants one month after the third dose in a 3-dose primary series with the immune response to all antigens induced by the same study vaccine outside Vietnam.
* To evaluate the immunogenicity of the study vaccine one month after the 3-dose primary series.
* To describe the persistence of all antibodies before receipt of the booster vaccination.
* To evaluate the immunogenicity of the study vaccine one month after the booster.

DETAILED DESCRIPTION:
Participants will receive a total of 5 doses of Hep B: One dose of Hep B monovalent vaccine given at birth or within 1 week after birth followed by 3 doses of the Sanofi Pasteur's hexavalent vaccine given as primary series at 2, 3, and 4 months of age and then a booster dose at 16 to 17 months of age, to comply with Vietnamese vaccination recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Aged 61 to 91 days on the day of the first study visit
* Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥2.5 kg
* Informed consent form has been signed and dated by the parent(s) or other legally acceptable representative (and by an independent witness if required by local regulations)
* Subject and parent/legally acceptable representative are able to attend all scheduled visits and to comply with all trial procedures
* Have received one dose of Hep B vaccine at birth or within 1 week after birth (documented according to the national recommendations).

Exclusion Criteria:

* Participation in the 4 weeks preceding the first trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination or planned receipt of any other vaccine within the period from 8 days before to 8 days after each subsequent trial vaccination except for Bacille Calmette Guerin (BCG) vaccination (any administration of oral poliovirus vaccine (OPV) in the context of oral poliovirus vaccine-national immunization days (NIDs) does not fall within the scope of this exclusion criterion)
* Previous vaccination against diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B (except the dose of Hep B vaccine given at birth or within 1 week after birth) diseases or Haemophilus influenzae type b infection with either the trial vaccine or another vaccine (any administration of OPV in the context of OPV-NIDs does not fall within the scope of this exclusion criterion)
* Past or current receipt of immune globulins, blood or blood-derived products or planned administration during the trial
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy since birth; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks since birth)
* History of diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B, or Haemophilus influenzae type b infections (confirmed either clinically, serologically or microbiologically)
* Known personal or maternal history of Human Immunodeficiency Virus (HIV), or hepatitis C seropositivity
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Known thrombocytopenia, as reported by the parent/legally acceptable representative
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* History of seizures
* In an emergency setting, or hospitalized involuntarily
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥38.0°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as a natural or adopted child of the Investigator, relatives or employee with direct involvement in the proposed study.

Ages: 61 Days to 91 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 354 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2017-01-11 (Actual); Study Completion 2017-01-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting Solicited Injection Site Reactions or Solicited Systemic Reactions | Within 7 days after vaccination
  Solicited injection site reactions: tenderness, erythema, and swelling (and extensive limb swelling for booster dose). Solicited systemic reactions: fever, vomiting, crying abnormal, drowsiness, appetite loss, and irritability

SECONDARY OUTCOMES:
Number of Subjects With Seroprotection/Seroconversion/Vaccine Response After Infant Series in Cohort 1 | Day 90 (1 month after third dose)
  Seroconversion:4-fold increase in anti-Pertussis(PT)& anti-Filamentous hemagglutinin(FHA) antibody(Ab) concentrations from pre-vaccination to one month after first dose.Vaccine response:anti-PT/anti-FHA Ab concentrations in Enzyme Linked Immunosorbent Assay(ELISA) units(EU)/mL>=4*Lower Limit of Quantitation(LLOQ) if pre-vaccination concentration <4*LLOQ/>=pre-vaccination concentration if prevaccination concentrations>=4*LLOQ. Seroprotection:anti-Diphtheria &anti-Tetanus>=0.01 International Units(IU)/mL&>=0.1 IU/mL;anti-PT &anti-FHA>=2 EU/mL &>=8 EU/mL;anti-Polyribosyl Ribitol Phosphate(PRP)>=0.15 microgram per milliliter(mcg/mL) &>=1.0mcg/mL;anti-Polio types 1,2,&3>=8(1/dilution),anti-Hepatitis B>=10 mili-international units per mililiter(mIU/mL)&>=100 mIU/mL
Number of Subjects With Seroprotection/Seroconversion/Vaccine and Booster Response Before and After Booster Vaccination in Cohort 1 | Day 425 (pre-booster) and Day 455 (1 month after booster dose)
  Seroconversion:4-fold increase in anti-PT & anti-FHA Ab concentrations from pre-booster vaccination to 1 month after booster dose.Vaccine response post-booster vaccination:post-booster Ab concentrations>=4*LLOQ if pre-dose 1 Ab concentrations<4*LLOQ/post-booster Ab concentrations>=predose 1 Ab concentrations if pre-dose 1>=4*LLOQ. Booster response:>=4 fold Ab concentrations increase from pre-dose 4 to one-month post-dose 4 if one-month post-dose 3<4*LLOQ/>=2 fold Ab concentrations increase from pre-dose 4 to one-month post-dose 4 if pre-dose 4>=4*LLOQ.Seroprotection:anti-Diphtheria
  & anti-Tetanus>=0.01 IU/mL &>=0.1 IU/mL &>=1.0 IU/mL;anti-PRP >=0.15 mcg/mL &>=1.0 mcg/mL;anti-Polio types 1, 2, & 3>=8 (1/dilution),anti-Hepatitis B>=10 mIU/mL &>=100 mIU/mL
Geometric Mean Titers or Geometric Mean Concentrations of DTaP-IPV-HB-PRP~T Antibodies Before and After Infant Series in Cohort | Day 90 (1 month after third dose)
  Geometric mean of concentrations of antibodies against PT, FHA, diphtheria, tetanus, PRP, poliovirus 1, 2 and 3, and Hep B
Geometric Mean Titers or Geometric Mean Concentrations of DTaP-IPV-HB-PRP~T Antibodies Before and After Booster Vaccination in Cohort 1 | Day 425 (pre-booster) and Day 455 (1 month after booster dose)
  Geometric mean of concentrations of antibodies against PT, FHA, diphtheria, tetanus, PRP, poliovirus 1, 2 and 3, and Hep B
Percentage of Subjects With Seroprotection/Seroconversion Rates after Infant Series in Cohort 1 and Group 3 of A3L15 (NCT01105559) | Day 90 (1 month after third dose)
  Seroconversion defined as 4-fold increase in anti-PT & anti-FHA Ab concentrations from pre-vaccination to one month after first dose. Seroprotection defined as following: anti-Diphtheria & anti-Tetanus >=0.01 IU/mL; anti-PT & anti-FHA >=4EU/mL; anti-PRP >=0.15 mcg/mL; anti-Polio types 1, 2, & 3 >=8 (1/dilution), anti-Hepatitis B >=10 mIU/mL. Results observed in Group 3 of Study A3L15 (NCT00362336), a study conducted in South Africa where participants had been given DTaP-IPV-HB-PRP~T at 6, 10, and 14 weeks of age following Hep B vaccination at birth, were used as the non-inferiority reference value

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (1):
- Preventive Medicine Centre of Thai Binh Province, Thái Bình, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com